CLINICAL TRIAL: NCT01986842
Title: The Impact of Habitual Dietary Protein Intake on the Anabolic Response in Elderly Men
Brief Title: Habitual Protein Intake and Muscle Protein Synthesis
Acronym: Pro-Hab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: METC 13-3-050
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Sarcopenia
Keywords: Muscle protein synthesis; Digestion and absorption kinetics; Leucine; Whey protein
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low protein (Experimental): Subject will receive a low protein diet (0.7 g/kg BW/day) for 14 days prior to the experimental trial
  Interventions: Dietary Supplement: Protein diet
- High protein (Experimental): Subjects will receive a high protein diet (1.5 g/kg BW/day) for 14 days prior to the experimental trial
  Interventions: Dietary Supplement: Protein diet

INTERVENTIONS:
Dietary Supplement: Protein diet — Subjects will receive either a low protein or a high protein diet for 14 days. High protein will be realized with protein supplements.

SUMMARY:
Protein intake stimulates muscle protein synthesis. From the standpoint of maintaining skeletal muscle mass with aging, it is important to optimize the adaptive response to food intake. However, a paucity of information is available describing the effects of habitual dietary protein intake (i.e. either high or low amounts of dietary protein consumed on a regular basis), on the subsequent meal-induced stimulation of muscle protein synthesis. An adaptation to a diet of several days or weeks may involve splanchnic and/or skeletal muscle adaptations that may further enhance, or decrease, the amino acid sensitivity of muscle protein synthesis after protein ingestion.

The aim of this study is to investigate the effect of a habitual (14 days) high protein diet when compared with low protein diet on digestion and absorption kinetics and the subsequent muscle protein synthetic response to dietary protein ingestion.

DETAILED DESCRIPTION:
During the adult life skeletal muscle mass remains fairly constant until the fourth or fifth decade. Then, the slow process of sarcopenia (the age-related loss of muscle mass) is believed to begin. The maintenance of skeletal muscle mass is regulated by a balance between the opposing processes of muscle protein synthesis and muscle protein breakdown. Food intake, dietary protein in particular, stimulates muscle protein synthesis and allows net muscle protein accretion throughout the day, which allows the normal maintenance of muscle mass in healthy individuals. Many studies have described the postprandial muscle protein synthetic response to protein intake and/or physical activity, and these acute findings have led to recommendations for protein intake for both athletes wishing to gain muscle mass as well as patients and elderly individuals to help them maintaining muscle mass. However, translating the acute findings from a single meal to long-term recommendations is perhaps premature, since scientists know very little with regard to how previous consumed meals affect the anabolic responsiveness to subsequent food intake. A characteristic of the adaptation to habitual high or low protein intake is thought to be associated with a change in the amplitude of diurnal cycle of whole body proteins. If this speculation is accurate, it implies that the muscle protein synthetic responses to feeding (differences between fasting and feeding muscle protein synthesis rates) are adapting to differing habitual protein intake, which may reduce (or enhance) the anabolic responsiveness to protein intake.

To gain a more complete scientific understanding, it is necessary to examine whether an adaptation does in fact occur after habitual high or low amounts of protein intake with regard to the anabolic response to subsequent protein intake. In the present investigation, we wish to investigate the impact of the habitual consumption of either high or low protein diets for 14 days on the anabolic responsiveness to a protein meal in healthy elderly. Previous work has determined that whole body adaptations to protein intake occur after >10 days. Collectively, our findings will be valuable to maximize the skeletal muscle adaptive response to food intake and, ultimately, to develop nutritional strategies for maintenance or enhancement of skeletal muscle mass in elderly men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age between 55 and 75 y
* BMI between 18.5 and 30 kg/m2

Exclusion Criteria:

* Lactose intolerance
* Smoking and alcohol abuse
* Diabetes
* Diagnosed GI tract diseases
* Arthritic conditions
* A history of neuromuscular problems
* Any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* Use of anticoagulants
* Participation in exercise program
* Hypertension, high blood pressure that is above 140/90 mmHg.

Ages: 55 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis rates | 0-5 h postprandial period
  Change in MPS rates during the postprandial phase when compared with the basal phase

SECONDARY OUTCOMES:
Digestion/Absorption kinetics | 0-5 h postprandial period
  Difference in digestion of the intrinsically labeled protein after a 14-day period of high vs. low protein diet

OTHER OUTCOMES:
Plasma insulin | 0-5 h postprandial period
Plasma amino acid concentrations | 0-5 h postprandial period
Whole-body protein metabolism | 0-5 h postprandial period
  Protein metabolism (breakdown, synthesis, oxidation, net balance)

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356
- [Derived] Gorissen SH, Horstman AM, Franssen R, Kouw IW, Wall BT, Burd NA, de Groot LC, van Loon LJ. Habituation to low or high protein intake does not modulate basal or postprandial muscle protein synthesis rates: a randomized trial. Am J Clin Nutr. 2017 Feb;105(2):332-342. doi: 10.3945/ajcn.115.129924. Epub 2016 Nov 30. PMID 27903518